CLINICAL TRIAL: NCT07396714
Title: Evaluation of the Efficacy & Safety of Topical Ivermectin Alone or in Combination With Microneedling as Novel Therapeutic Options for Cutaneous Non-genital Warts Versus Topical Salicylic Acid ؛ Randomized Controlled Clinical Trial.
Brief Title: the Efficacy of Ivermectin Alone or With Microneedling in Treatment of Cutaneous Warts.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Sayed Abdelaziz, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ivermectin for cutaneous warts
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Warts
Keywords: topical ivermectin with microneedling in warts treatment
MeSH Terms: conditions — Warts | interventions — Ivermectin; Percutaneous Collagen Induction; Salicylic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- topical ivermectin (Experimental)
  Interventions: Drug: Ivermectin
- microneedling (Experimental): patients with cutaneous warts will be treated with microneedling.
  Interventions: Device: microneedling
- microneedling with ivermectin (Experimental): patients with cutaneous warts will be treated with topical ivermectin with microneedling.
  Interventions: Drug: Ivermectin; Device: microneedling
- topical salicylic acid (Active Comparator): patients with cutaneous warts will be treated with topical salicylic acid.
  Interventions: Drug: Salicylic Acid

INTERVENTIONS:
Drug: Ivermectin — patients with non-genital cutaneous warts will be treated by topical application of ivermectin : topical ivermectin 1% will be applied under occlusion overnight daily then revaluated every 2 weeks for maximum 12 weeks
  Arms: microneedling with ivermectin; topical ivermectin
Device: microneedling — patients with non-genital cutaneous warts will be treated by microneedling (2mm depth) every 2-weeks until complete clearance or for a maximum of 12weeks
  Arms: microneedling; microneedling with ivermectin
Drug: Salicylic Acid — patients with non-genital cutaneous warts will be treated by topical application of ivermectin : cotton soaked with topical salicylic acid will be applied under occlusion overnight daily then revaluated every 2 weeks for maximum 12 weeks
  Arms: topical salicylic acid

SUMMARY:
To compare between the efficacy and safety of topical ivermectin alone, microneedling with topical ivermectin and topical salicylic acid in treatment of cutaneous warts.

topical ivermectin 1% will be applied on warts whole night clinical assessment will be done every 2 weeks

Microneedling will be performed on the lesion using a microneedling pen type device with a 1-cm tip diameter at a 2-mm depth setting for 2-3 minutes until pinpoint bleebing occurs 1 mL of topical ivermectin 1% will be applied on to the wart tissue.

Sessions: Sessions will be performed every 2 weeks until complete cure or for maximum 6 sessions (total 3 month)

DETAILED DESCRIPTION:
Wart is a benign skin growth caused by infection with the human papillomavirus (HPV). These lesions typically appear as rough, raised projections on the skin, often on the hands, feet, or other areas. More than 200 types of HPV have been identified.

Worldwide, warts (due to HPV) are extremely common. Estimates suggest about 7-12% of the global population have cutaneous warts at any given time, and among school-aged children the prevalence can reach 10-20%.

The main types of cutaneous non genital warts are : Common warts, often appears on hands &fingers ,Plantar warts: occur on the soles of the feet, Flat warts occur often on the face, legs.

Warts cause pain (especially plantar types), cosmetic embarrassment, in addition to risk of transmission to others There are several therapeutic modalities for warts: include destructive agents (keratolytics, cryotherapy, curettage and cautery, laser, photodynamic therapy), antimitotic agents (podophyllin, bleomycin, retinoids), immune stimulants (topical sensitizers, cimetidine), and topical virucidal agents (formaldehyde, glutaraldehyde) No single treatment is effective in most of patients, available options often painful ,associated with recurrence and have risks like scarring or infection.

Ivermectin, which is traditionally used as an anti- helminthic agent, has been found to have a range of effects beyond its initial well known anti-parasitic use, that include: immune modulatory, anti-viral and anti- proliferative effect. The immune modulatory effect of Ivermectin depends on it's ability to modulate pro-inflammatory cytokines. It also has antiviral role by inhibition of viral replication, several studies have addressed its antiviral activity against a diverse range of viruses, leading to its exploration for use in treating SARS-CoV-2 during the most recent global pandemic .

Emerging literature highlights the potential use of ivermectin as a promising candidate for anticancer therapy through inhibition of the proliferation of the tumour cells by regulating multiple signalling pathways.

In dermatology topical ivermectin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of hair lice & rosacea.

The anti-proliferative & antiviral activity of ivermectin suggests it's use in the treatment of HPV infection. Oral ivermectin demonstrated efficacy in a case study for treatment of resistant cutaneous warts, 10 patients clinically diagnosed cutaneous warts were enrolled. Each patient received oral ivermectin at a dose of 200 μg/kg body weight once daily for 3 weeks .Results indicated a substantial reduction in the number and size of warts in 8 patients, 4 patients of them experienced complete resolution of their warts. The efficacy of topical ivermectin in treatment of cutaneous warts still uncovered.

Microneedling is also an effective treatment option for HPV by Immune activation: Micro-injuries initiate a localized inflammatory and wound-healing response, which can enhance the immune system's ability to recognize and clear human papillomavirus (HPV)-infected cells. It also enhance drug penetration: When paired with topical agents (e.g., bleomycin, 5 fluorouracil, methotrexate), microneedling facilitates deeper and more uniform penetration into the wart tissue. This increases drug effectiveness while potentially reducing systemic side effects.

This study will be conducted to explore the potential efficacy of topical ivermectin 1% either alone or in combination with assist delivery via microneedling in treatment of non genital cutaneous warts.

ELIGIBILITY:
Inclusion Criteria:

* patients with cutaneous non genital warts aged 11:80 y.
* No concurrent systemic or topical treatment of warts

Exclusion Criteria:

* Genital warts.

  * Pregnancy and lactation.
  * History of any bleeding, clotting disorder or using anticoagulants
  * Chronic systemic diseases such as chronic renal failure, hepaticinsufficiency, and cardiovascular disorders.
  * patients who received any treatment for warts in the last month before the study.
  * Patients with history of neuropathy or peripheral ischemia.
  * Patients with signs of inflammation or infection.
  * Patients with history of a serious systemic or anaphylactic reaction or allergy to ivermectin.

Ages: 11 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the efficacy of topical ivermectin in treatment of cutaneous warts. | baseline
  clinical assessment of warts at the baseline & each visit comparing photographs at different timeline .

SECONDARY OUTCOMES:
evaluation of the efficacy of topical ivermectin combined with microneedling in treatment of cutaneous warts. | baseline
  clinical assessment of warts at the baseline & at each visit every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alaa mohamed ghazaly, MD, Study Director — Assiut University; Ayman Mohamed Mahran, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehta N. Case study of oral ivermectin in patients with cutaneous warts. J Cardiovasc Dis Res. 2024;15(12):6438-46
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30406683/